CLINICAL TRIAL: NCT01920347
Title: Prospective Pilot Trial to Evaluate the NeurOptics Pupillometer and Clinical Examination of the Pupillary Reflex After Cardiac Arrest
Brief Title: The Neurological Pupil Index (NPi) on Intensive Care Unit (ICU) Trial
Acronym: NPI-ON-ICU
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, C. Storm, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: 112823
Record Dates: First submitted 2013-05-27; First posted 2013-08-12 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Hypoxic Encephalopathy
Keywords: hypoxic encephalopathy; cardiac arrest; outcome; pupillary reflex
MeSH Terms: conditions — Hypoxia, Brain; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neurological Pupil index: The NPi will be measured during treatment

SUMMARY:
The trial will evaluate the use of the "Neurological Pupil index" NPi, measured with the digital pupillometer (NeurOptics) compared to clinical examination for better reliability. The investigators hypothesize that digital evaluation will offer a higher sensitivity/ specificity compared to clinical examination.

DETAILED DESCRIPTION:
Absent pupillary reaction after cardiac arrest might indicate a severe hypoxic encephalopathy. Because the examination of the pupillary reaction is easy it is part of the clinical routine but due to the different medication and the dynamic process of reperfusion injury to the brain a clinical evaluation might be not precise enough. The NPi has been shown to be superior to clinical evaluation in different settings but without regard towards cardiac arrest survivors. The Pupillometer is a hand-held, cordless, and simple to use device which removes subjectivity in the measurement of pupil size and the pupillary light reflex.

ELIGIBILITY:
Inclusion Criteria:

* all survivors after cardiac arrest

Exclusion Criteria:

* underlying disease limiting the pupillary reflex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Survivors after cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Neurological Pupil index (NPi) on a scale from 0-5 | up to 7 days
  NPi values by the device on a scale by 0-5; >3 indicates normal reaction; <3 abnormal.

SECONDARY OUTCOMES:
Cerebral performance category (CPC) | Patients will be followed for the duration of hospital stay, an expected average of 2 weeks
  cerebral performance category; 1-2 good outcome; 3-5 poor outcome

CONTACTS AND LOCATIONS:
Overall Officials: Christian Storm, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (2):
- Germany (2):
  - Charité Universitätsmedizin Berlin, Berlin
  - Charité Universitätsmedizin, Berlin